CLINICAL TRIAL: NCT04200482
Title: Testing a Scalable Nutrition and Physical Activity Program for Breast Cancer Survivors: A Dose-Finding Pilot Study
Brief Title: Lifestyle Program (Scalable Nutrition and Physical Activity) for the Improvement of Nutrition and Physical Activity in Stage 0-III Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1006427; NCI-2019-07643 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10335 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
Keywords: Breast Cancer Survivors; Diet; eHealth; Nutrition; Physical Activity; Breast
MeSH Terms: conditions — Breast Carcinoma In Situ; Motor Activity | interventions — Behavior Therapy; Health; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (low dose nutrition and PA class, eHealth intervention) (Active Comparator): Participants attend one diet and physical activity class delivered remotely via Zoom and receive an eHealth communication intervention for 6 months.
  Interventions: Behavioral: One Diet and Physical Activity Session; Other: Electronic (e) Health (eHealth) Communication Intervention; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm B (high dose nutrition and PA class, eHealth intervention) (Experimental): Participants attend 12 twice monthly diet and physical activity online sessions delivered remotely via Zoom and receive an eHealth communication intervention for 6 months.
  Interventions: Other: Electronic (e) Health (eHealth) Communication Intervention; Behavioral: Twelve Diet and Physical Activity Group Sessions; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Behavioral: One Diet and Physical Activity Session — Attend 1 remote diet and physical activity session
  Other Names: Behavior or Lifestyle Modifications; behavior modification; Behavior Conditioning Therapy; Behavioral Interventions; Behavioral Treatments
  Arms: Arm A (low dose nutrition and PA class, eHealth intervention)
Other: Electronic (e) Health (eHealth) Communication Intervention — Receive eHealth communication intervention
Behavioral: Twelve Diet and Physical Activity Group Sessions — Attend 12 remote diet and physical activity sessions in 6 months
  Other Names: Behavior or Lifestyle Modifications; behavior modification; Behavior Conditioning Therapy; Behavioral Interventions; Behavioral Treatments
  Arms: Arm B (high dose nutrition and PA class, eHealth intervention)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
The purpose of this phase II trial is to identify the most effective dose level (number of classes) of a diet and physical activity lifestyle program based on how well it improves diet and physical activity in stage 0-III breast cancer survivors. Study results may provide researchers with information on how to best implement diet and physical activity recommendations among breast cancer survivors.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A (LOW DOSE): Participants attend one diet and physical activity class delivered remotely via Zoom and receive an eHealth communication intervention for 6 months.

ARM B (HIGH DOSE): Participants attend 12 twice monthly diet and physical activity online sessions delivered remotely via Zoom and receive an eHealth communication intervention for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of stage 0-III breast cancer in the past 10 years at the time of enrollment
* No evidence of recurrent or metastatic disease
* No uncontrolled diabetes mellitus defined as glycosylated hemoglobin (Hgb A1C) > 8%
* No uncontrolled hypertension per Seattle Cancer Care Alliance (SCCA) standard of care
* At least 60 days post final chemotherapy, biologic therapy, or radiation therapy and/or surgery. Current use of endocrine therapy is permitted (e.g., tamoxifen and aromatase inhibitors)
* Access to phone for study contacts
* Access to smartphone, tablet, or computer and internet to attend online session(s) and receive study electronic eHealth communication (text messages and access to website)
* Willing and able to attend the online session(s) on Saturdays, or via online accessed videos, for up to 12 sessions in 6 months
* Successfully complete all run-in activities, including at-home and over the phone assessments, 7 days of collecting physical activity data via accelerometer, and providing blood and stool sample
* Willing and able to complete all study activities for 6 months after randomization
* Participants must consume < 5 servings of fruits and vegetables per day and/or engage in < 150 minutes per week of moderate to vigorous physical activity, as assessed by brief questionnaires
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Scale of performance status score of 0 or 1 for performance status.
* Signed physician approval for diet change and physical activity
* Able to understand and willing to sign written informed electronic (e) consent in English

Exclusion Criteria:

* Participants must not be active smokers within the past 30 days.
* Women must not be pregnant at time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Accrual rate | At 6 months
  Accrual rate will be measured by number of participants randomized during each month of study accrual.
Adherence: Session(s) Attendance | At 6 months
  Adherence will be measured by number of online session(s) attended per participant.
Adherence: Responsiveness to eHealth communication | At 6 months
  Adherence will be measured by the number of responses to text messages per participant.
Biospecimen collection rate | At 6 months
  Biospecimen collection rate will be assessed based on number of biospecimens collected.
Retention | At 6 months
  Retention will be measured by the number of completed study assessments per participants.
Acceptability: Questions during exit interview | At 6 months
  Acceptability will be measured by questions asking about trial acceptability in the exit questionnaire.

SECONDARY OUTCOMES:
Change in daily servings of fruits and vegetables per day | Baseline to 6 months
  Will be assessed by 24-hour dietary recalls.
Change in minutes per week of moderate-to-vigorous physical activity | Baseline to 6 months
  Will be assessed by 7-day accelerometer data.
Change in systemic inflammation | Baseline to 6 months
  Will be assessed by fasting blood concentrations of high sensitivity C-reactive protein.
Change in gut barrier permeability | Baseline to 6 months
  Will be assessed by fasting circulating levels of gut bacterial endotoxin liposaccharide-binding protein.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Davidson, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium; Heather Greenlee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ueland K, Sanchez SC, Rillamas-Sun E, Shen H, Schattenkerk L, Garcia G, VanDoren M, Myers SA, Santiago-Torres M, Di C, Dey N, Guthrie KA, Yung R, Davidson NE, Greenlee H. A digital health intervention to improve nutrition and physical activity in breast cancer survivors: Rationale and design of the Cook and Move for Your Life pilot and feasibility randomized controlled trial. Contemp Clin Trials. 2022 Dec;123:106993. doi: 10.1016/j.cct.2022.106993. Epub 2022 Nov 3. PMID 36336249
- [Derived] Rillamas-Sun E, Schattenkerk L, Cobos S, Ueland K, Gaffney AO, Greenlee H. Characteristics of Users of the Cook for Your Life Website, an Online Nutrition Resource for Persons Affected by Cancer: Descriptive Study. JMIR Cancer. 2022 Jul 5;8(3):e37212. doi: 10.2196/37212. PMID 35788100

DOCUMENTS (1):
  • Informed Consent Form (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT04200482/ICF_000.pdf